CLINICAL TRIAL: NCT06038968
Title: Anatomical and Functional Outcomes of Use of Methotrexate Infusion and Intrasilicone Injection During Diabetic Vitrectomy
Brief Title: Methotrexate Infusion and Intrasilicone Injection During Diabetic Vitrectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Abdallah Mohsen Mohamed Safwat, assistant lecturer, ophthalmology department, faculty of medicine, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MTX DM vitrectomy
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Retinopathy; Vitreomacular Traction
Keywords: Methotrexate; proliferative diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate group (Experimental): methotrexate group will receive 40 mg of MTX in 500 ml of irrigation fluid during vitrectomy and 250 ug intra-silicone oil injection at the end of vitrectomy
  Interventions: Drug: Methotrexate 25 MG/ML; Procedure: parsplana vitrectomy
- Control group (Placebo Comparator): control group will not receive MTX in irrigation fluid during vitrectomy nor intra-silicone at the end of vitrectomy
  Interventions: Procedure: parsplana vitrectomy

INTERVENTIONS:
Drug: Methotrexate 25 MG/ML — Methotrexate is a folate derivative that inhibits several enzymes responsible for nucleotide synthesis. This inhibition leads to suppression of inflammation as well as prevention of cell division.
  Other Names: Methotrexate Mylan 50 mg/2 mL
  Arms: Methotrexate group
Procedure: parsplana vitrectomy — Pars plana vitrectomy (PPV) is a technique in vitreoretinal surgery that enables access to the posterior segment for treating tractional retinal detachment in advanced proliferative diabetic retinopathy, in a controlled, closed system.

SUMMARY:
The goal of this interventional clinical trial is to assess anatomical and functional outcomes of methotrexate use in irrigating fluid during parsplana vitrectomy combined with intrasilicone injection at end of surgery in patients with advanced proliferative diabetic retinopathy.

The main questions it aims to answer are:

1. Does methotrexate use in irrigating fluid during parsplana vitrectomy combined with intrasilicone injection at end of surgery decrease the post operative vitreoretinal proliferation after vitrectomy in patients with advanced proliferative diabetic retinopathy?
2. Does methotrexate use in irrigating fluid during parsplana vitrectomy combined with intrasilicone injection at end of surgery improve post operative functional outcome after vitrectomy in patients with advanced proliferative diabetic retinopathy?

Researchers will compare the anatomical and functional outcomes after vitrectomy in patients with advanced proliferative diabetic retinopathy without using methotrexate.

DETAILED DESCRIPTION:
Tractional macular detachment (TMD) or macula threatening tractional retinal detachment (TRD) and combined tractional-rhegmatogenous retinal detachment (TRD/RRD) are considered as important indications for vitreoretinal intervention.

Although a growing number of eyes with TMD and TRD/RRD are successfully treated with a single procedure, retinal re-detachment associated with fibrovascular proliferation or proliferative vitreoretinopathy (PVR) is still a major cause of failure of the surgery.

Previous studies have shown increased expression of inflammatory cytokines and growth factors in both proliferative diabetic retinopathy (PDR) and PVR.

Methotrexate (MTX) is an anti-neoplastic and anti-inflammatory agent used to treat a variety of malignancies and rheumatologic diseases.

In ophthalmology, systemic and intraocular MTX has been successfully used for indeterminate uveitis, sarcoid uveitis and intraocular lymphoma.

MTX has been recently found to inhibit PVR by stopping cellular proliferation and promoting organized apoptosis. MTX has also been found to be effective in lowering the incidence of PVR when used as an adjunct in irrigation fluid during vitrectomy for retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

- Patients with diabetic tractional macular detachment or combined tractional- rhegmatogenous retinal detachment

Exclusion Criteria:

* Previous vitreoretinal surgery.
* Pregnant or lactating female.
* Co-existing pathology that might induce PVR such as penetrating ocular trauma or uveitis, co-existing congenital anomalies or hereditary vitreoretinopathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
assess retinal layers by optical coherence tomography | one month after pars plana vitrectomy and one month after silicone oil evacuation
  presence of epiretinal membrane, cystic changes in retina, central macular thickens
assess functional outcomes by multifocal electroretinogram | one month after pars plana vitrectomy and one month after silicone oil evacuation
  latency and amplitude of main P wave

SECONDARY OUTCOMES:
Anterior segment slit lamp biomicroscopic examination | one month after pars plana vitrectomy
  assess anterior segment inflammation as iritis or posterior synechia
visual acuity | one month after pars plana vitrectomy and one month after silicone oil evacuation
  by logMAR (Logarithm of the Minimum Angle of Resolution)

CONTACTS AND LOCATIONS:
Overall Officials: Rabie MM Hasanin, Professor, Study Chair — ophthalmology department, faculty of medicine, Minia university hospital; Khaled MS morad, Professor, Study Director — ophthalmology department, faculty of medicine, Minia university hospital; Ahmed MA Shawkat, Professor, Study Director — ophthalmology department, faculty of medicine, Minia university hospital; Mohamed Tarek AM Mostafa, Ass. Prof., Study Director — ophthalmology department, faculty of medicine, Minia university hospital
Locations (1):
- ophthalmology department, Minia university hospital, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
email the main investigator for requested data

REFERENCES:
- [Background] Newman DK. Surgical management of the late complications of proliferative diabetic retinopathy. Eye (Lond). 2010 Mar;24(3):441-9. doi: 10.1038/eye.2009.325. Epub 2010 Feb 5. PMID 20139916
- [Background] Meleth AD, Carvounis PE. Outcomes of vitrectomy for tractional retinal detachment in diabetic retinopathy. Int Ophthalmol Clin. 2014 Spring;54(2):127-39. doi: 10.1097/IIO.0000000000000021. No abstract available. PMID 24613889
- [Background] Gologorsky D, Thanos A, Vavvas D. Therapeutic interventions against inflammatory and angiogenic mediators in proliferative diabetic retinopathy. Mediators Inflamm. 2012;2012:629452. doi: 10.1155/2012/629452. Epub 2012 Sep 17. PMID 23028203
- [Background] Zhou J, Wang S, Xia X. Role of intravitreal inflammatory cytokines and angiogenic factors in proliferative diabetic retinopathy. Curr Eye Res. 2012 May;37(5):416-20. doi: 10.3109/02713683.2012.661114. Epub 2012 Mar 12. PMID 22409294
- [Background] Ricker LJ, Kijlstra A, Kessels AG, de Jager W, Liem AT, Hendrikse F, La Heij EC. Interleukin and growth factor levels in subretinal fluid in rhegmatogenous retinal detachment: a case-control study. PLoS One. 2011 Apr 27;6(4):e19141. doi: 10.1371/journal.pone.0019141. PMID 21556354
- [Background] Samson CM, Waheed N, Baltatzis S, Foster CS. Methotrexate therapy for chronic noninfectious uveitis: analysis of a case series of 160 patients. Ophthalmology. 2001 Jun;108(6):1134-9. doi: 10.1016/s0161-6420(01)00576-0. PMID 11382642
- [Background] Smith JR, Rosenbaum JT, Wilson DJ, Doolittle ND, Siegal T, Neuwelt EA, Pe'er J. Role of intravitreal methotrexate in the management of primary central nervous system lymphoma with ocular involvement. Ophthalmology. 2002 Sep;109(9):1709-16. doi: 10.1016/s0161-6420(02)01125-9. PMID 12208721
- [Background] Amarnani D, Machuca-Parra AI, Wong LL, Marko CK, Stefater JA, Stryjewski TP, Eliott D, Arboleda-Velasquez JF, Kim LA. Effect of Methotrexate on an In Vitro Patient-Derived Model of Proliferative Vitreoretinopathy. Invest Ophthalmol Vis Sci. 2017 Aug 1;58(10):3940-3949. doi: 10.1167/iovs.16-20912. PMID 28777835